CLINICAL TRIAL: NCT00929110
Title: A 52-week Treatment, Randomized, Double-blind, Placebo-controlled, With Open-label Tiotropium, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Glycopyrronium Bromide (NVA237) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: 1-year Study to Assess the Efficacy, Safety, and Tolerability of Glycopyrronium Bromide (NVA237) in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: GLOW2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNVA237A2303; 2008-008394-63 (EudraCT Number)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; NVA237; glycopyrronium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Glycopyrronium bromide 50 μg (Experimental): Patients inhaled glycopyrronium bromide 50 μg once daily in the morning between 8:00 AM and 10:00 AM via a single-dose dry-powder inhaler (SDDPI) for 52 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Glycopyrronium bromide
- Placebo to glycopyrronium bromide (Placebo Comparator): Patients inhaled placebo to glycopyrronium bromide once daily in the morning between 8:00 AM and 10:00 AM via a single-dose dry-powder inhaler (SDDPI) for 52 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to glycopyrronium bromide
- Tiotropium 18 μg (Active Comparator): Patients inhaled tiotropium 18 μg once daily in the morning between 8:00 AM and 10:00 AM via a single-dose dry-powder inhaler (SDDPI) for 52 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Glycopyrronium bromide — Glycopyrronium bromide was supplied in powder-filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Other Names: NVA237
  Arms: Glycopyrronium bromide 50 μg
Drug: Placebo to glycopyrronium bromide — Placebo to glycopyrronium bromide was supplied in powder-filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Placebo to glycopyrronium bromide
Drug: Tiotropium — Tiotropium was supplied in powder-filled capsules together with the Handihaler® device.
  Arms: Tiotropium 18 μg

SUMMARY:
This study was designed to investigate the 1 year efficacy and safety of the 50 µg once daily (od) dose of glycopyrronium bromide (NVA237) in patients with moderate to severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged ≥ 40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure.
2. Patients with moderate to severe stable chronic obstructive pulmonary disease (COPD, Stage II or Stage III) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines 2008.
3. Current or ex-smokers who have a smoking history of at least 10 pack years.
4. Patients with a post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 30% and < 80% of the predicted normal, and post-bronchodilator FEV1/forced vital capacity (FVC) < 0.7 at Visit 2 (Day -14).
5. Patients, according to daily electronic diary data between Visit 2 (Day -14) and Visit 3 (Day 1), with a total score of 1 or more on at least 4 of the last 7 days prior to Visit 3 (Day 1).

Exclusion Criteria:

1. Pregnant women or nursing mothers (pregnancy confirmed by positive urine pregnancy test).
2. Women of child-bearing potential, unless using an approved method of medical or surgical contraception.
3. Patients requiring long term oxygen therapy (> 15 h a day) on a daily basis for chronic hypoxemia, or who have been hospitalized for an exacerbation of their airways disease in the 6 weeks prior to Visit 1 (Day -21) or between Visit 1 (Day -21) and Visit 3 (Day 1).
4. Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1 (Day -21).
5. Patients who, in the judgment of the investigator or the responsible Novartis personnel, have a clinically relevant laboratory abnormality or a clinically significant condition.
6. Patients with any history of asthma indicated by (but not limited to) a blood eosinophil count > 600/mm^3 (at Visit 1, Day -21) and onset of symptoms prior to age 40 years.
7. Patients with a history of long QT syndrome or whose QTc measured at Visit 1 (Day -21) (Fridericia method) is prolonged (> 450 ms for males or > 470 ms for females.

Other protocol-defined inclusion/exclusion criteria may apply to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1066 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (135):
- United States (71):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Montgomery, Alabama
  - Novartis Investigator Site, Fort Smith, Arkansas
  - Novartis Investigator Site, Anaheim, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Lakewood, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site, Mission Viejo, California
  - Novartis Investigator Site, Paramount, California
  - Novartis Investigator Site, Riverside, California
  - Novartis Investigative Site, Rolling Hills Estates, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, Colorado Springs, Colorado
  - Novartis Investigative site, DeLand, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Miami Beach, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Panama City, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigator Site, Winter Park, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Blue Ridge, Georgia
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigator Site, Coeur d'Alene, Idaho
  - Novartis Investigator Site, Skokie, Illinois
  - Novartis Investigator Site, New Albany, Indiana
  - Novartis Investigator Site, Valparaiso, Indiana
  - Novartis Investigator Site, Council Bluffs, Iowa
  - Novartis Investigator Site, Iowa City, Iowa
  - Novartis Investigator Site, Shawnee, Kansas
  - Novartis Investigative Center, Crescent Springs, Kentucky
  - Novartis Investigative Site, Crestview Hills, Kentucky
  - Novartis Investigative Site, Hazard, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigator Site, Lafayette, Louisiana
  - Novartis Investigator Site, Sunset, Louisiana
  - Novartis Investigator Site, Boys Town, Maine
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Taunton, Massachusetts
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Bozeman, Montana
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Papillion, Nebraska
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Endwell, New York
  - Novartis Investigative site, Charlotte, North Carolina
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigator Site, Sylvania, Ohio
  - Novartis Investigator Site, Toledo, Ohio
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Medford, Oregon
  - Novartis Investigator Site, Portland, Oregon
  - Novartis Investigative Site, Downingtown, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, East Providence, Rhode Island
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigator Site, Austin, Texas
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigator Site, New Braunfels, Texas
  - Novartis Investigator Site, San Antonio, Texas
  - Novartis Investigator Site, Provo, Utah
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigator Site, Tacoma, Washington
  - Novartis Investigator Site, Milwaukee, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, La Plata - Bueno Aire
  - Novartis Investigative Site, Parana Entre Rios
  - Novartis Investigative Site, Rosario
  - Novartis Investigative Site, San Miguel de Tucumán
- Canada (8):
  - Novartis Investigator Site, Brampton
  - Novartis Investigator Site, Calgary
  - Novartis Investigator Site, Edmonton
  - Novartis Investigator Site, Kelowna
  - Novartis Investigator Site, Langley
  - Novartis Investigator Site, Niagara Falls
  - Novartis Investigator Site, Québec
  - Novartis Investigator Site, Ste-Foy
- Chile (3):
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Talcahuano
  - Novartis Investigative Site, Viña del Mar
- France (3):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, München
- Hungary (2):
  - Novartis Investigative Site, Gyonsyos
  - Novartis Investigative Site, Siokok
- Israel (5):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Rehovot
- Italy (3):
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Parma
- Mexico (3):
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigative Site, Monterrey
  - Novartis Investigative Site, San Luis Potosí City
- Novartis Investigative Site, Sneek, Netherlands
- New Zealand (5):
  - Novartis Investigator Site, Auckland
  - Novartis Investigator Site, Christchurch
  - Novartis Investigator Site, Hamilton
  - Novartis Investigator Site, Tauranga
  - Novartis Investigator Site, Wellington
- Peru (2):
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Santiago de Surco
- Poland (9):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bystra
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Piekary Slaskic
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Warsaw
- Russia (6):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Yaroslavl
- South Korea (4):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gyeonggi-go
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul

REFERENCES:
- [Derived] D'Urzo A, Kerwin E, Overend T, D'Andrea P, Chen H, Goyal P. Once daily glycopyrronium for the treatment of COPD: pooled analysis of the GLOW1 and GLOW2 studies. Curr Med Res Opin. 2014 Mar;30(3):493-508. doi: 10.1185/03007995.2013.858618. Epub 2013 Nov 19. PMID 24156566
- [Derived] Kerwin E, Hebert J, Gallagher N, Martin C, Overend T, Alagappan VK, Lu Y, Banerji D. Efficacy and safety of NVA237 versus placebo and tiotropium in patients with COPD: the GLOW2 study. Eur Respir J. 2012 Nov;40(5):1106-14. doi: 10.1183/09031936.00040712. Epub 2012 Jul 26. PMID 23060624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1993 patients were screened from 180 participating sites, of whom 1066 were randomized to 1 of the 3 treatment groups in a 2:1:1 ratio glycopyrronium bromide:placebo:tiotropium.
Period: Overall Study
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Started | 529 | 269 | 268
Completed | 411 | 193 | 206
Not Completed | 118 | 76 | 62
Not completed — Adverse Event | 40 | 29 | 18
Not completed — Subject withdrew consent | 40 | 23 | 26
Not completed — Unsatisfactory therapeutic effect | 20 | 9 | 6
Not completed — Lost to Follow-up | 7 | 7 | 3
Not completed — Protocol deviation | 5 | 2 | 4
Not completed — Administrative problems | 4 | 1 | 2
Not completed — Death | 2 | 2 | 2
Not completed — Abnormal laboratory value(s) | 0 | 1 | 0
Not completed — Abnormal test procedure result(s) | 0 | 1 | 1
Not completed — Patient inability to use the device | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg | Total
Number analyzed (Participants) | 525 | 268 | 267 | 1060
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are based on the safety population which was defined as all patients who received at least 1 dose of study medication whether they were randomized or not. The number of patients in the safety population was less than the number of randomized patients, ie, some randomized patients did not receive study medication (4 in the glycopyrronium bromide group, 1 in the placebo group, and 1 in the tiotropium group).
  years | 63.5 (9.05) | 63.6 (9.14) | 63.9 (8.25) | 63.6 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data are based on the safety population which was defined as all patients who received at least 1 dose of study medication whether they were randomized or not. The number of patients in the safety population was less than the number of randomized patients, ie, some randomized patients did not receive study medication (4 in the glycopyrronium bromide group, 1 in the placebo group, and 1 in the tiotropium group).
  Participants
    Female | 186 | 95 | 99 | 380
    Male | 339 | 173 | 168 | 680

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 15 minutes and 23 hours 45 minutes post-dose. The analysis included baseline FEV1 measurement, baseline inhaled corticosteroid use (Yes/No), FEV1 prior to inhalation of short-acting β2 agonist (SABA), and FEV1 45 min post-inhalation of SABA as covariates.
Time Frame: Week 12
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 513 | 245 | 253
Liters | 1.469 (0.0141) | 1.372 (0.0173) | 1.455 (0.0170)

2. Secondary Outcome: Transition Dyspnea Index (TDI) at Week 26
Description: The TDI measured changes in dyspnea from baseline during treatment and included 3 domains: Functional impairment (activities of daily living), magnitude of task (intensity of activity), and magnitude of effort (difficulty breathing). Each domain was rated from -3 to 3 (major deterioration-major improvement). The total score ranged from -9 to 9; minus scores indicate deterioration. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: Week 26
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 470 | 217 | 238
Units on a scale | 2.13 (0.240) | 1.32 (0.289) | 2.26 (0.281)

3. Secondary Outcome: Health-related Quality of Life (QoL) Assessed With the St. George Respiratory Questionnaire (SGRQ) at Week 52
Description: The SGRQ contained 51 patient-rated items divided into three components: Symptoms (respiratory symptoms, their frequency, and severity), Activity (activities that cause or are limited by breathlessness), and Impacts (social functioning and psychological disturbances resulting from airway disease). A total score for the 3 components was calculated and ranged from 0 to 100. Higher values indicate greater impairment of QoL. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 499 | 248 | 251
Units on a scale | 40.85 (0.854) | 44.16 (1.040) | 41.32 (1.024)

4. Secondary Outcome: Time to First Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation During the Study (Baseline to Week 52)
Description: Time to first moderate or severe COPD exacerbation was calculated as the number of days from baseline to the day on which the patient experienced the first moderate or severe COPD exacerbation. A COPD exacerbation was considered to be moderate if treatment with systemic corticosteroids and/or antibiotic was required. A COPD exacerbation was considered to be severe if treatment for moderate severity and hospitalization was required.
Time Frame: Baseline to Week 52 (patients with no moderate or severe exacerbations who completed the study were censored at the final visit date, which may have exceeded 52 weeks)
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 525 | 268 | 267
Days | 363.0 [1 to 402] | 231.0 [1 to 380] | 364.0 [1 to 423]

5. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication Taken During the Study (Baseline to Week 52)
Description: The number of puffs of rescue medication taken in the previous 12 hours was recorded in the Patient Diary in the morning and evening. The mean daily number of puffs of rescue medication taken was calculated by dividing the number of puffs of rescue medication per day over the 52 weeks of the study by the number of days with non-missing rescue medication data. Rescue medication data recorded during the 14 day run-in period was used to calculate the baseline. The analysis included the same covariates as the primary Outcome Measure. A positive change score indicates more puffs taken.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 523 | 263 | 263
Puffs | -1.58 (0.151) | -1.20 (0.184) | -1.83 (0.183)

6. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 1, Week 26, and Week 52
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 15 minutes and 23 hours 45 minutes post-dose. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: Day 1, Week 26, and Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 500 | 250 | 245
Liters
  Day 1 | 1.478 (0.0088) | 1.388 (0.0109) | 1.471 (0.0109)
  Week 26 (n=451, 219, 233) | 1.458 (0.0161) | 1.324 (0.0196) | 1.408 (0.0191)
  Week 52 (n=416, 196, 210) | 1.412 (0.0157) | 1.303 (0.0198) | 1.392 (0.0191)

7. Secondary Outcome: Trough Forced Vital Capacity (FVC) at Day 1, Week 12, Week 26, and Week 52
Description: Trough FVC is defined as the average of the post-dose 23 h 15 min and the 23 h 45 min FVC values. Just prior to FVC measurement, patients performed normal tidal breathing. The patient was given a few breaths warning before being told "At the end of the next normal breath out, take a deep breath all the way in"; they were then verbally encouraged to make a maximal effort before relaxing. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: Day 1, Week 12, Week 26, and Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 500 | 250 | 245
Liters
  Day 1 | 2.936 (0.0165) | 2.757 (0.0205) | 2.930 (0.0206)
  Week 12 (n=442, 204, 217) | 2.985 (0.0265) | 2.802 (0.0329) | 2.970 (0.0323)
  Week 26 (n=418, 196, 208) | 2.962 (0.0299) | 2.758 (0.0361) | 2.892 (0.0355)
  Week 52 (n=395, 186, 201) | 2.866 (0.0335) | 2.687 (0.0399) | 2.866 (0.0383)

8. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 5, 15, and 30 Minutes; 1, 2, 3, 4, 6, 8, 10, and 12 Hours; 23 Hours 15 Minutes; and 23 Hours 45 Minutes Post-dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The analysis included the same covariates as the primary Outcome Measure. Data was not collected at all time points for all Days and Weeks.
Time Frame: 5, 15, and 30 minutes; 1, 2, 3, 4, 6, 8, 10, and 12 hours; 23 hours 15 minutes; and 23 hours 45 minutes post-dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Population: Full Analysis Set (FAS), serial spirometry subgroup: A subgroup of approximately one third of all randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 144 | 79 | 76
Liters
  Day 1, minute 5 (n=135, 74, 74) | 1.494 (0.0135) | 1.416 (0.0166) | 1.447 (0.0164)
  Day 1, minute 15 (n=139, 75, 74) | 1.548 (0.0152) | 1.428 (0.0185) | 1.485 (0.0185)
  Day 1, minute 30 (n=143, 77, 74) | 1.561 (0.0180) | 1.409 (0.0218) | 1.483 (0.0219)
  Day 1, hour 1 (n=144, 76, 75) | 1.583 (0.0172) | 1.404 (0.0213) | 1.514 (0.0212)
  Day 1, hour 2 (n=144, 75, 75) | 1.639 (0.0202) | 1.445 (0.0248) | 1.569 (0.0247)
  Day 1, hour 3 (n=143, 74, 73) | 1.629 (0.0199) | 1.435 (0.0249) | 1.587 (0.0248)
  Day 1, hour 4 (n=144, 70, 74) | 1.599 (0.0221) | 1.415 (0.0281) | 1.560 (0.0275)
  Day 1, hour 6 (n=142, 71, 74) | 1.578 (0.0204) | 1.426 (0.0255) | 1.575 (0.0252)
  Day 1, hour 8 (n=137, 70, 75) | 1.544 (0.0226) | 1.431 (0.0284) | 1.545 (0.0278)
  Day1, hour 10 (n=134, 72, 75) | 1.546 (0.0235) | 1.415 (0.0290) | 1.537 (0.0286)
  Day 1, hour 12 (n=130, 69, 70) | 1.522 (0.0254) | 1.369 (0.0307) | 1.480 (0.0306)
  Day 1, hour 23, minute 15 (n=129, 71, 72) | 1.471 (0.0214) | 1.396 (0.0259) | 1.481 (0.0255)
  Day 1, hour 23, minute 45 (n=128, 74, 75) | 1.518 (0.0210) | 1.446 (0.0252) | 1.499 (0.0249)
  Day 15, minute 5 (n=135, 65, 73) | 1.494 (0.0246) | 1.421 (0.0315) | 1.490 (0.0299)
  Day 15, minute 15 (n=133, 70, 72) | 1.530 (0.0246) | 1.411 (0.0307) | 1.537 (0.0303)
  Day 15, minute 30 (n= 139, 70, 74) | 1.551 (0.0236) | 1.417 (0.0297) | 1.516 (0.0289)
  Day 15, hour 1 (n=140, 68, 74) | 1.575 (0.0242) | 1.409 (0.0305) | 1.540 (0.0296)
  Week 5, minute 5 (n=134, 66, 68) | 1.550 (0.0247) | 1.448 (0.0319) | 1.525 (0.0305)
  Week 5, minute 15 (n=136, 67, 70) | 1.575 (0.0239) | 1.452 (0.0305) | 1.543 (0.0295)
  Week 5, minute 30 (n=135, 67, 70) | 1.630 (0.0260) | 1.481 (0.0327) | 1.584 (0.0317)
  Week 9, minute 5 (n=128, 66, 70) | 1.562 (0.0268) | 1.417 (0.0341) | 1.520 (0.0326)
  Week 9, minute 15 (n=130, 66, 71) | 1.583 (0.0267) | 1.441 (0.0340) | 1.534 (0.0326)
  Week 9, minute 30 (n=130, 67, 71) | 1.603 (0.0265) | 1.427 (0.0335) | 1.549 (0.0323)
  Week 12, minute 5 (n=130, 69, 70) | 1.497 (0.0254) | 1.385 (0.0319) | 1.474 (0.0315)
  Week 12, minute 15 (n=129, 67, 66) | 1.523 (0.0251) | 1.373 (0.0317) | 1.481 (0.0315)
  Week 12, minute 30 (n=133, 69, 67) | 1.517 (0.0275) | 1.362 (0.0336) | 1.488 (0.0335)
  Week 12, hour 1 (n=132, 67, 69) | 1.557 (0.0273) | 1.369 (0.0341) | 1.519 (0.0333)
  Week 12, hour 2 (n=129, 65, 68) | 1.596 (0.0290) | 1.434 (0.0365) | 1.565 (0.0353)
  Week 12, hour 3 (n=126, 64, 69) | 1.600 (0.0291) | 1.443 (0.0375) | 1.566 (0.0353)
  Week 12, hour 4 (n=124, 64, 68) | 1.584 (0.0319) | 1.442 (0.0407) | 1.535 (0.0383)
  Week 12, hour 6 (n=123, 63, 69) | 1.558 (0.0321) | 1.443 (0.0407) | 1.520 (0.0381)
  Week 12, hour 8 (n=121, 64, 69) | 1.535 (0.0310) | 1.408 (0.0385) | 1.479 (0.0374)
  Week 12, hour 10 (n=124, 61, 69) | 1.541 (0.0296) | 1.435 (0.0392) | 1.532 (0.0365)
  Week 12, hour 12 (n=122, 58, 68) | 1.522 (0.0313) | 1.422 (0.0417) | 1.487 (0.0382)
  Week 12, hour 16 (n=109, 56, 57) | 1.431 (0.0320) | 1.360 (0.0425) | 1.378 (0.0404)
  Week 12, hour 22 (n=117, 60, 63) | 1.420 (0.0268) | 1.349 (0.0350) | 1.371 (0.0333)
  Week 12, hour 23, minute 15 (n=126, 66, 67) | 1.518 (0.0269) | 1.456 (0.0345) | 1.520 (0.0335)
  Week 12, hour 23, minute 45 (n=124, 65, 63) | 1.513 (0.0294) | 1.470 (0.0377) | 1.488 (0.0374)
  Week 16, minute 5 (n=123, 65, 64) | 1.538 (0.0296) | 1.430 (0.0362) | 1.515 (0.0359)
  Week 16, minute 15 (n=124, 65, 65) | 1.557 (0.0309) | 1.422 (0.0380) | 1.530 (0.0377)
  Week 16, minute 30 (n=125, 65, 65) | 1.570 (0.0303) | 1.409 (0.0370) | 1.535 (0.0368)
  Week 20, minute 5 (n=125, 66, 63) | 1.518 (0.0281) | 1.393 (0.0348) | 1.453 (0.0351)
  Week 20, minute 15 (n=124, 65, 63) | 1.535 (0.0285) | 1.380 (0.0354) | 1.479 (0.0356)
  Week 20, minute 30 (n=125, 65, 63) | 1.576 (0.0277) | 1.391 (0.0349) | 1.502 (0.0350)
  Week 26, minute 5 (n=123, 62, 64) | 1.483 (0.0278) | 1.361 (0.0368) | 1.415 (0.0352)
  Week 26, minute 15 (n=121, 61, 61) | 1.521 (0.0280) | 1.377 (0.0373) | 1.464 (0.0358)
  Week 26, minute 30 (n=125, 64, 64) | 1.529 (0.0285) | 1.353 (0.0372) | 1.439 (0.0359)
  Week 26, hour 1 (n=127, 64, 64) | 1.546 (0.0275) | 1.364 (0.0359) | 1.462 (0.0349)
  Week 26, hour 2 (n=124, 64, 63) | 1.590 (0.0317) | 1.422 (0.0403) | 1.520 (0.0395)
  Week 26, hour 3 (n=124, 64, 64) | 1.614 (0.0303) | 1.442 (0.0391) | 1.555 (0.0380)
  Week 26, hour 4 (n=124, 64, 62) | 1.577 (0.0304) | 1.416 (0.0384) | 1.519 (0.0377)
  Week 26, hour 23, minute 15 (n=120, 55, 61) | 1.477 (0.0323) | 1.374 (0.0422) | 1.416 (0.0399)
  Week 26, hour 23, minute 45 (n=117, 56, 61) | 1.483 (0.0296) | 1.401 (0.0395) | 1.405 (0.0376)
  Week 34, minute 5 (n=125, 62, 63) | 1.515 (0.0293) | 1.359 (0.0385) | 1.407 (0.0372)
  Week 34, minute 15 (n=123, 62, 63) | 1.529 (0.0300) | 1.360 (0.0394) | 1.425 (0.0379)
  Week 34, minute 30 (n=125, 62, 62) | 1.567 (0.0302) | 1.353 (0.0398) | 1.452 (0.0385)
  Week 34, hour 1 (n=125, 62, 63) | 1.557 (0.0285) | 1.352 (0.0376) | 1.472 (0.0361)
  Week 42, minute 5 (n=119, 61, 58) | 1.512 (0.0305) | 1.394 (0.0401) | 1.490 (0.0394)
  Week 42, minute 15 (n=123, 61, 58) | 1.520 (0.0305) | 1.412 (0.0403) | 1.491 (0.0396)
  Week 42, minute 30 (n=123, 61, 58) | 1.537 (0.0332) | 1.391 (0.0431) | 1.517 (0.0424)
  Week 50, minute 5 (n=120, 60, 57) | 1.490 (0.0269) | 1.357 (0.0348) | 1.422 (0.0341)
  Week 50, minute 15 (n=123, 60, 57) | 1.529 (0.0285) | 1.375 (0.0369) | 1.452 (0.0362)
  Week 50, minute 30 (n=123, 60, 58) | 1.545 (0.0287) | 1.368 (0.0375) | 1.470 (0.0366)
  Week 52, minute 5 (n=124, 60, 57) | 1.456 (0.0276) | 1.337 (0.0368) | 1.377 (0.0359)
  Week 52, minute 15 (n=122, 59, 58) | 1.502 (0.0282) | 1.380 (0.0378) | 1.428 (0.0364)
  Week 52, minute 30 (n=125, 62, 58) | 1.483 (0.0280) | 1.366 (0.0370) | 1.407 (0.0362)
  Week 52, hour 1 (n=125, 62, 57) | 1.525 (0.0271) | 1.356 (0.0359) | 1.439 (0.0352)
  Week 52, hour 2 (n=124, 61, 58) | 1.554 (0.0295) | 1.418 (0.0393) | 1.479 (0.0382)
  Week 52, hour 3 (n=123, 62, 56) | 1.558 (0.0263) | 1.384 (0.0349) | 1.487 (0.0345)
  Week 52, hour 4 (n=121, 60, 55) | 1.535 (0.0297) | 1.381 (0.0395) | 1.468 (0.0390)
  Week 52, hour 6 (n=118, 59, 54) | 1.494 (0.0294) | 1.370 (0.0392) | 1.461 (0.0388)
  Week 52, hour 8 (n=119, 59, 54) | 1.473 (0.0300) | 1.358 (0.0398) | 1.418 (0.0394)
  Week 52, hour 10 (n=119, 59, 55) | 1.478 (0.0304) | 1.349 (0.0397) | 1.419 (0.0391)
  Week 52, hour 12 (n=120, 58, 52) | 1.451 (0.0334) | 1.369 (0.0446) | 1.347 (0.0444)
  Week 52, hour 16 (n=117, 53, 46) | 1.377 (0.0309) | 1.277 (0.0422) | 1.329 (0.0420)
  Week 52, hour 22 (n=118, 60, 52) | 1.391 (0.0302) | 1.314 (0.0397) | 1.282 (0.0396)
  Week 52, hour 23, 15 minutes (n=121, 62, 57) | 1.447 (0.0287) | 1.362 (0.0378) | 1.387 (0.0371)
  Week 52, hour 23, 45 minutes (n=122, 61, 57) | 1.434 (0.0281) | 1.337 (0.0372) | 1.359 (0.0364)

9. Secondary Outcome: Forced Vital Capacity (FVC) 5, 15, and 30 Minutes; 1, 2, 3, 4, 6, 8, 10, and 12 Hours; 23 Hours 15 Minutes; and 23 Hours 45 Minutes Post-dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Description: Just prior to FVC measurement, patients performed normal tidal breathing. The patient was given a few breaths warning before being told "At the end of the next normal breath out, take a deep breath all the way in"; they were then verbally encouraged to make a maximal effort before relaxing. The analysis included the same covariates as the primary Outcome Measure. Data was not collected at all time points for all Days and Weeks.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 144 | 79 | 76
Liters
  Day 1, minute 5 (n=135, 74, 74) | 3.027 (0.0304) | 2.826 (0.0363) | 2.956 (0.0363)
  Day 1, minute 15 (n=139, 75, 74) | 3.050 (0.0335) | 2.802 (0.0403) | 2.991 (0.0406)
  Day 1, minute 30 (n=143, 77, 74) | 3.055 (0.0343) | 2.752 (0.0416) | 2.979 (0.0422)
  Day 1, hour 1 (n=144, 76, 75) | 3.148 (0.0377) | 2.791 (0.0460) | 3.041 (0.0463)
  Day 1, hour 2 (n=144, 75, 75) | 3.179 (0.0373) | 2.802 (0.0460) | 3.049 (0.0461)
  Day 1, hour 3 (n=143, 74, 73) | 3.190 (0.0433) | 2.826 (0.0526) | 3.119 (0.0531)
  Day 1, hour 4 (n=144, 70, 74) | 3.138 (0.0414) | 2.783 (0.0515) | 3.102 (0.0512)
  Day 1, hour 6 (n=142, 71, 74) | 3.173 (0.0419) | 2.846 (0.0514) | 3.148 (0.0513)
  Day 1, hour 8 (n=137, 70, 75) | 3.071 (0.0404) | 2.804 (0.0506) | 3.074 (0.0498)
  Day1, hour 10 (n=134, 72, 75) | 3.134 (0.0414) | 2.865 (0.0514) | 3.119 (0.0510)
  Day 1, hour 12 (n=130, 69, 70) | 3.030 (0.0444) | 2.709 (0.0535) | 3.012 (0.0537)
  Day 1, hour 23, minute 15 (n=129, 71, 72) | 2.991 (0.0385) | 2.800 (0.0478) | 2.988 (0.0471)
  Day 1, hour 23, minute 45 (n=128, 74, 75) | 3.014 (0.0364) | 2.817 (0.0444) | 2.994 (0.0442)
  Day 15, minute 5 (n=135, 65, 73) | 3.051 (0.0439) | 2.793 (0.0553) | 3.014 (0.0534)
  Day 15, minute 15 (n=133, 70, 72) | 3.103 (0.0443) | 2.790 (0.0536) | 3.103 (0.0536)
  Day 15, minute 30 (n= 139, 70, 74) | 3.134 (0.0420) | 2.825 (0.0519) | 3.078 (0.0513)
  Day 15, hour 1 (n=140, 68, 74) | 3.152 (0.0434) | 2.770 (0.0537) | 3.060 (0.0528)
  Week 5, minute 5 (n=134, 66, 68) | 3.139 (0.0430) | 2.866 (0.0551) | 3.071 (0.0534)
  Week 5, minute 15 (n=136, 67, 70) | 3.165 (0.0501) | 2.850 (0.0611) | 3.092 (0.0602)
  Week 5, minute 30 (n=135, 67, 70) | 3.248 (0.0540) | 2.884 (0.0644) | 3.180 (0.0636)
  Week 9, minute 5 (n=128, 66, 70) | 3.195 (0.0543) | 2.826 (0.0644) | 3.097 (0.0632)
  Week 9, minute 15 (n=130, 66, 71) | 3.167 (0.0507) | 2.823 (0.0615) | 3.101 (0.0603)
  Week 9, minute 30 (n=130, 67, 71) | 3.231 (0.0567) | 2.821 (0.0675) | 3.149 (0.0664)
  Week 12, minute 5 (n=130, 69, 70) | 3.060 (0.0492) | 2.728 (0.0596) | 3.023 (0.0596)
  Week 12, minute 15 (n=129, 67, 66) | 3.081 (0.0482) | 2.740 (0.0588) | 3.018 (0.0593)
  Week 12, minute 30 (n=133, 69, 67) | 3.058 (0.0479) | 2.696 (0.0585) | 3.027 (0.0591)
  Week 12, hour 1 (n=132, 67, 69) | 3.164 (0.0543) | 2.737 (0.0663) | 3.098 (0.0655)
  Week 12, hour 2 (n=129, 65, 68) | 3.190 (0.0526) | 2.784 (0.0664) | 3.155 (0.0649)
  Week 12, hour 3 (n=126, 64, 69) | 3.240 (0.0569) | 2.864 (0.0713) | 3.146 (0.0685)
  Week 12, hour 4 (n=124, 64, 68) | 3.119 (0.0576) | 2.745 (0.0714) | 3.084 (0.0686)
  Week 12, hour 6 (n=123, 63, 69) | 3.158 (0.0594) | 2.852 (0.0731) | 3.120 (0.0700)
  Week 12, hour 8 (n=121, 64, 69) | 3.083 (0.0534) | 2.760 (0.0657) | 3.011 (0.0644)
  Week 12, hour 10 (n=124, 61, 69) | 3.130 (0.0581) | 2.860 (0.0722) | 3.117 (0.0692)
  Week 12, hour 12 (n=122, 58, 68) | 3.072 (0.0599) | 2.771 (0.0770) | 3.020 (0.0722)
  Week 12, hour 16 (n=109, 56, 57) | 2.933 (0.0645) | 2.701 (0.0800) | 2.880 (0.0785)
  Week 12, hour 22 (n=117, 60, 63) | 2.924 (0.0517) | 2.673 (0.0647) | 2.870 (0.0629)
  Week 12, hour 23, minute 15 (n=126, 66, 67) | 3.091 (0.0548) | 2.862 (0.0676) | 3.110 (0.0671)
  Week 12, hour 23, minute 45 (n=124, 65, 63) | 3.055 (0.0507) | 2.826 (0.0630) | 3.004 (0.0638)
  Week 16, minute 5 (n=123, 65, 64) | 3.156 (0.0608) | 2.864 (0.0719) | 3.104 (0.0723)
  Week 16, minute 15 (n=124, 65, 65) | 3.156 (0.0576) | 2.801 (0.0695) | 3.082 (0.0699)
  Week 16, minute 30 (n=125, 65, 65) | 3.198 (0.0552) | 2.815 (0.0676) | 3.112 (0.0679)
  Week 20, minute 5 (n=125, 66, 63) | 3.093 (0.0526) | 2.781 (0.0630) | 2.993 (0.0643)
  Week 20, minute 15 (n=124, 65, 63) | 3.112 (0.0545) | 2.770 (0.0655) | 3.029 (0.0666)
  Week 20, minute 30 (n=125, 65, 63) | 3.157 (0.0559) | 2.778 (0.0677) | 3.050 (0.0688)
  Week 26, minute 5 (n=123, 62, 64) | 2.994 (0.0528) | 2.700 (0.0670) | 2.954 (0.0658)
  Week 26, minute 15 (n=121, 61, 61) | 3.041 (0.0513) | 2.692 (0.0652) | 2.976 (0.0644)
  Week 26, minute 30 (n=125, 64, 64) | 3.054 (0.0464) | 2.700 (0.0597) | 2.994 (0.0589)
  Week 26, hour 1 (n=127, 64, 64) | 3.077 (0.0520) | 2.678 (0.0658) | 3.016 (0.0651)
  Week 26, hour 2 (n=124, 64, 63) | 3.110 (0.0516) | 2.771 (0.0655) | 3.080 (0.0650)
  Week 26, hour 3 (n=124, 64, 64) | 3.210 (0.0648) | 2.871 (0.0765) | 3.176 (0.0762)
  Week 26, hour 4 (n=124, 64, 62) | 3.111 (0.0551) | 2.791 (0.0664) | 3.086 (0.0664)
  Week 26, hour 23, minute 15 (n=120, 55, 61) | 3.056 (0.0600) | 2.803 (0.0749) | 2.932 (0.0721)
  Week 26, hour 23, minute 45 (n=117, 56, 61) | 2.998 (0.0512) | 2.752 (0.0667) | 2.895 (0.0646)
  Week 34, minute 5 (n=125, 62, 63) | 3.023 (0.0573) | 2.731 (0.0715) | 2.881 (0.0706)
  Week 34, minute 15 (n=123, 62, 63) | 3.016 (0.0553) | 2.731 (0.0691) | 2.898 (0.0683)
  Week 34, minute 30 (n=125, 62, 62) | 3.081 (0.0555) | 2.687 (0.0715) | 2.971 (0.0708)
  Week 34, hour 1 (n=125, 62, 63) | 3.072 (0.0564) | 2.703 (0.0707) | 2.963 (0.0699)
  Week 42, minute 5 (n=119, 61, 58) | 3.033 (0.0583) | 2.716 (0.0744) | 3.069 (0.0746)
  Week 42, minute 15 (n=123, 61, 58) | 3.022 (0.0539) | 2.695 (0.0706) | 3.065 (0.0699)
  Week 42, minute 30 (n=123, 61, 58) | 3.057 (0.0565) | 2.723 (0.0734) | 3.098 (0.0734)
  Week 50, minute 5 (n=120, 60, 57) | 3.022 (0.0596) | 2.731 (0.0727) | 2.963 (0.0726)
  Week 50, minute 15 (n=123, 60, 57) | 3.042 (0.0592) | 2.702 (0.0726) | 2.937 (0.0725)
  Week 50, minute 30 (n=123, 60, 58) | 3.094 (0.0613) | 2.731 (0.0749) | 2.985 (0.0747)
  Week 52, minute 5 (n=124, 60, 57) | 2.940 (0.0551) | 2.645 (0.0701) | 2.860 (0.0702)
  Week 52, minute 15 (n=122, 59, 58) | 2.960 (0.0518) | 2.640 (0.0675) | 2.935 (0.0666)
  Week 52, minute 30 (n=125, 62, 58) | 2.939 (0.0499) | 2.625 (0.0650) | 2.929 (0.0652)
  Week 52, hour 1 (n=125, 62, 57) | 3.031 (0.0564) | 2.617 (0.0698) | 2.980 (0.0704)
  Week 52, hour 2 (n=124, 61, 58) | 3.062 (0.0556) | 2.714 (0.0689) | 3.021 (0.0689)
  Week 52, hour 3 (n=123, 62, 56) | 3.108 (0.0648) | 2.716 (0.0766) | 3.053 (0.0779)
  Week 52, hour 4 (n=121, 60, 55) | 3.021 (0.0585) | 2.694 (0.0724) | 2.978 (0.0735)
  Week 52, hour 6 (n=118, 59, 54) | 2.986 (0.0614) | 2.690 (0.0770) | 2.982 (0.0781)
  Week 52, hour 8 (n=119, 59, 54) | 2.961 (0.0646) | 2.637 (0.0793) | 2.942 (0.0805)
  Week 52, hour 10 (n=119, 59, 55) | 3.000 (0.0701) | 2.687 (0.0840) | 3.012 (0.0844)
  Week 52, hour 12 (n=120, 58, 52) | 2.881 (0.0631) | 2.636 (0.0831) | 2.849 (0.0847)
  Week 52, hour 16 (n=117, 53, 46) | 2.857 (0.0694) | 2.542 (0.0857) | 2.772 (0.0873)
  Week 52, hour 22 (n=118, 60, 52) | 2.812 (0.0670) | 2.604 (0.0810) | 2.716 (0.0827)
  Week 52, hour 23, 15 minutes (n=121, 62, 57) | 2.888 (0.0595) | 2.678 (0.0751) | 2.852 (0.0755)
  Week 52, hour 23, 45 minutes (n=122, 61, 57) | 2.855 (0.0558) | 2.607 (0.0700) | 2.797 (0.0702)

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 5, 15, and 30 Minutes; and 1, 2, 3, and 4 Hours Post Dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Description: as for outcome 8
Time Frame: 5, 15, and 30 minutes; and 1, 2, 3, 4 hours post-dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 525 | 268 | 267
Liters
  Day 1, minute 5 (n=495, 255, 253) | 1.443 (0.0067) | 1.357 (0.0081) | 1.402 (0.0081)
  Day 1, minute 15 (n=502, 255, 254) | 1.501 (0.0074) | 1.359 (0.0090) | 1.437 (0.0090)
  Day 1, minute 30 (n=507, 252, 254) | 1.524 (0.0103) | 1.357 (0.0126) | 1.468 (0.0125)
  Day 1, hour 1 (n=511, 256, 254) | 1.552 (0.0082) | 1.353 (0.0101) | 1.484 (0.0101)
  Day 1, hour 2 (n=513, 253, 252) | 1.612 (0.0090) | 1.397 (0.0113) | 1.549 (0.0112)
  Day 1, hour 3 (n=510, 248, 252) | 1.590 (0.0088) | 1.389 (0.0111) | 1.560 (0.0109)
  Day 1, hour 4 (n=504, 239, 250) | 1.590 (0.0095) | 1.396 (0.0121) | 1.549 (0.0117)
  Day 1, hour 23, minute 15 (n=481, 243, 239) | 1.459 (0.0093) | 1.364 (0.0115) | 1.457 (0.0115)
  Day 1, hour 23, minute 45 (n=474, 239, 232) | 1.482 (0.0094) | 1.390 (0.0117) | 1.473 (0.0118)
  Day 15, minute 5 (n=498, 223, 243) | 1.491 (0.0123) | 1.368 (0.0157) | 1.472 (0.0151)
  Day 15, minute 15 (n=487, 229, 239) | 1.527 (0.0123) | 1.371 (0.0154) | 1.514 (0.0151)
  Day 15, minute 30 (n=503, 233, 242) | 1.538 (0.0122) | 1.368 (0.0152) | 1.504 (0.0150)
  Day 15, hour 1 (n=501, 229, 240) | 1.561 (0.0121) | 1.379 (0.0153) | 1.525 (0.0150)
  Week 5, minute 5 (n=476, 221, 231) | 1.509 (0.0125) | 1.371 (0.0161) | 1.488 (0.0157)
  Week 5, minute 15 (n=479, 222, 234) | 1.538 (0.0126) | 1.389 (0.0162) | 1.508 (0.0157)
  Week 5, minute 30 (n=480, 223, 234) | 1.564 (0.0129) | 1.396 (0.0165) | 1.525 (0.0160)
  Week 9, minute 5 (n=454, 217, 227) | 1.529 (0.0126) | 1.366 (0.0159) | 1.499 (0.0157)
  Week 9, minute 15 (n=459, 220, 225) | 1.550 (0.0132) | 1.376 (0.0164) | 1.515 (0.0163)
  Week 9, minute 30 (n=460, 220, 226) | 1.569 (0.0125) | 1.378 (0.0158) | 1.531 (0.0157)
  Week 12, minute 5 (n=453, 212, 230) | 1.502 (0.0136) | 1.349 (0.0173) | 1.477 (0.0167)
  Week 12, minute 15 (n=448, 205, 222) | 1.527 (0.0131) | 1.352 (0.0171) | 1.501 (0.0166)
  Week 12, minute 30 (n=455, 212, 226) | 1.522 (0.0139) | 1.352 (0.0176) | 1.491 (0.0170)
  Week 12, hour 1 (n=455, 210, 227) | 1.556 (0.0139) | 1.364 (0.0178) | 1.528 (0.0171)
  Week 12, hour 2 (n=446, 207, 225) | 1.595 (0.0145) | 1.423 (0.0185) | 1.558 (0.0178)
  Week 12, hour 3 (n=444, 204, 225) | 1.592 (0.0145) | 1.414 (0.0186) | 1.561 (0.0177)
  Week 12, hour 4 (n=437, 202, 224) | 1.558 (0.0152) | 1.416 (0.0193) | 1.534 (0.0183)
  Week 12, hour 23, minute 15 (n=430, 200, 214) | 1.481 (0.0143) | 1.381 (0.0183) | 1.457 (0.0177)
  Week 12, hour 23, minute 45 (n=426, 195, 205) | 1.493 (0.0149) | 1.413 (0.0190) | 1.472 (0.0187)
  Week 16, minute 5 (n=429, 207, 218) | 1.514 (0.0151) | 1.373 (0.0185) | 1.487 (0.0181)
  Week 16, minute 15 (n=428, 209, 219) | 1.530 (0.0155) | 1.372 (0.0189) | 1.491 (0.0186)
  Week 16, minute 30 (n=433, 209, 220) | 1.546 (0.0160) | 1.372 (0.0194) | 1.505 (0.0190)
  Week 20, minute 5 (n=430, 206, 218) | 1.495 (0.0159) | 1.351 (0.0198) | 1.464 (0.0192)
  Week 20, minute 15 (n=430, 207, 220) | 1.525 (0.0164) | 1.362 (0.0203) | 1.495 (0.0196)
  Week 20, minute 30 (n=431, 207, 221) | 1.544 (0.0164) | 1.362 (0.0203) | 1.498 (0.0195)
  Week 26, minute 5 (421, 202, 213) | 1.479 (0.0153) | 1.339 (0.0189) | 1.429 (0.0185)
  Week 26, minute 15 (n=414, 200, 207) | 1.504 (0.0155) | 1.340 (0.0193) | 1.458 (0.0191)
  Week 26, minute 30 (n=424, 206, 213) | 1.513 (0.0161) | 1.341 (0.0196) | 1.451 (0.0193)
  Week 26, hour 1 (n=425, 206, 212) | 1.541 (0.0160) | 1.345 (0.0193) | 1.487 (0.0190)
  Week 26, hour 2 (n=420, 203, 208) | 1.570 (0.0176) | 1.388 (0.0212) | 1.524 (0.0210)
  Week 26, hour 3 (n=416, 204, 213) | 1.570 (0.0181) | 1.398 (0.0216) | 1.526 (0.0211)
  Week 26, hour 4 (n=416, 203, 208) | 1.547 (0.0175) | 1.384 (0.0211) | 1.504 (0.0208)
  Week 26, hour 23, minute 15 (n=405, 187, 202) | 1.464 (0.0175) | 1.326 (0.0217) | 1.415 (0.0212)
  Week 26, hour 23, minute 45 (n=401, 185, 198) | 1.474 (0.0175) | 1.354 (0.0218) | 1.426 (0.0215)
  Week 34, minute 5 (n=408, 194, 212) | 1.481 (0.0167) | 1.338 (0.0210) | 1.422 (0.0202)
  Week 34, minute 15 (n=407, 191, 214) | 1.508 (0.0172) | 1.333 (0.0215) | 1.443 (0.0206)
  Week 34, minute 30 (n=410, 196, 215) | 1.518 (0.0172) | 1.331 (0.0214) | 1.444 (0.0206)
  Week 34, hour 1 (n=412, 195, 215) | 1.534 (0.0171) | 1.331 (0.0213) | 1.464 (0.0205)
  Week 42, minute 5 (n=398, 189, 199) | 1.489 (0.0172) | 1.342 (0.0218) | 1.459 (0.0213)
  Week 42, minute 15 (n=405, 188, 201) | 1.511 (0.0171) | 1.344 (0.0218) | 1.477 (0.0211)
  Week 42, minute 30 (n=405, 189, 201) | 1.518 (0.0183) | 1.350 (0.0229) | 1.496 (0.0222)
  Week 50, minute 5 (n=386, 185, 199) | 1.454 (0.0155) | 1.336 (0.0197) | 1.429 (0.0190)
  Week 50, minute 15 (n=391, 187, 203) | 1.496 (0.0156) | 1.341 (0.0199) | 1.462 (0.0192)
  Week 50, minute 30 (n=392, 186, 204) | 1.504 (0.0166) | 1.341 (0.0210) | 1.475 (0.0200)
  Week 52, minute 5 (n=401, 188, 197) | 1.436 (0.0155) | 1.305 (0.0200) | 1.419 (0.0195)
  Week 52, minute 15 (n=394, 183, 200) | 1.471 (0.0159) | 1.323 (0.0208) | 1.451 (0.0198)
  Week 52, minute 30 (n=402, 189, 202) | 1.471 (0.0164) | 1.319 (0.0209) | 1.451 (0.0202)
  Week 52, hour 1 (n=404, 190, 201) | 1.499 (0.0161) | 1.325 (0.0205) | 1.482 (0.0198)
  Week 52, hour 2 (n=402, 186, 202) | 1.526 (0.0177) | 1.363 (0.0224) | 1.511 (0.0214)
  Week 52, hour 3 (n=400, 186, 199) | 1.525 (0.0171) | 1.344 (0.0215) | 1.509 (0.0207)
  Week 52, hour 4 (n=397, 184, 199) | 1.504 (0.0176) | 1.346 (0.0222) | 1.501 (0.0213)
  Week 52, hour 23, minute 15 (n=388, 183, 198) | 1.419 (0.0169) | 1.303 (0.0215) | 1.397 (0.0205)
  Week 52, hour 23, minute 45 (n=395, 185, 199) | 1.424 (0.0165) | 1.320 (0.0210) | 1.411 (0.0201)

11. Secondary Outcome: Forced Vital Capacity (FVC) 5, 15, and 30 Minutes; and 1, 2, 3, and 4 Hours Post-dose at Days 1 and 15; and Weeks 5, 9, 12, 16, 20, 26, 34, 42, 50, and 52
Description: as for outcome 9
Time Frame: as for outcome 10
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 525 | 268 | 267
Liters
  Day 1, minute 5 (n=495, 255, 253) | 2.915 (0.0145) | 2.731 (0.0174) | 2.856 (0.0174)
  Day 1, minute 15 (n=502, 255, 254) | 2.982 (0.0164) | 2.719 (0.0199) | 2.903 (0.0198)
  Day 1, minute 30 (n=507, 252, 254) | 3.004 (0.0177) | 2.692 (0.0219) | 2.937 (0.0217)
  Day 1, hour 1 (n=511, 256, 254) | 3.074 (0.0173) | 2.732 (0.0214) | 2.975 (0.0213)
  Day 1, hour 2 (n=513, 253, 252) | 3.119 (0.0182) | 2.762 (0.0227) | 3.033 (0.0226)
  Day 1, hour 3 (n=510, 248, 252) | 3.129 (0.0193) | 2.811 (0.0243) | 3.073 (0.0239)
  Day 1, hour 4 (n=504, 239, 250) | 3.076 (0.0192) | 2.767 (0.0244) | 3.031 (0.0237)
  Day 1, hour 23, minute 15 (n=481, 243, 239) | 2.926 (0.0178) | 2.745 (0.0220) | 2.923 (0.0220)
  Day 1, hour 23, minute 45 (n=474, 239, 232) | 2.930 (0.0178) | 2.749 (0.0221) | 2.923 (0.0224)
  Day 15, minute 5 (n=498, 223, 243) | 2.984 (0.0222) | 2.760 (0.0282) | 2.980 (0.0272)
  Day 15, minute 15 (n=487, 229, 239) | 3.016 (0.0220) | 2.748 (0.0274) | 3.030 (0.0270)
  Day 15, minute 30 (n=503, 233, 242) | 3.028 (0.0212) | 2.756 (0.0269) | 3.018 (0.0265)
  Day 15, hour 1 (n=501, 229, 240) | 3.068 (0.0213) | 2.757 (0.0271) | 3.023 (0.0267)
  Week 5, minute 5 (n=476, 221, 231) | 3.004 (0.0215) | 2.768 (0.0277) | 3.011 (0.0270)
  Week 5, minute 15 (n=479, 222, 234) | 3.024 (0.0234) | 2.771 (0.0294) | 3.024 (0.0286)
  Week 5, minute 30 (n=480, 223, 234) | 3.085 (0.0243) | 2.804 (0.0305) | 3.063 (0.0297)
  Week 9, minute 5 (n=454, 217, 227) | 3.047 (0.0262) | 2.767 (0.0313) | 3.029 (0.0309)
  Week 9, minute 15 (n=459, 220, 225) | 3.050 (0.0257) | 2.764 (0.0312) | 3.046 (0.0311)
  Week 9, minute 30 (n=460, 220, 226) | 3.079 (0.0265) | 2.768 (0.0322) | 3.079 (0.0319)
  Week 12, minute 5 (n=453, 212, 230) | 2.991 (0.0253) | 2.726 (0.0313) | 2.978 (0.0304)
  Week 12, minute 15 (n=448, 205, 222) | 3.003 (0.0252) | 2.735 (0.0316) | 3.004 (0.0307)
  Week 12, minute 30 (n=455, 212, 226) | 2.985 (0.0251) | 2.707 (0.0314) | 2.987 (0.0306)
  Week 12, hour 1 (n=455, 210, 227) | 3.062 (0.0267) | 2.741 (0.0333) | 3.048 (0.0322)
  Week 12, hour 2 (n=446, 207, 225) | 3.093 (0.0266) | 2.801 (0.0335) | 3.065 (0.0324)
  Week 12, hour 3 (n=444, 204, 225) | 3.129 (0.0275) | 2.839 (0.0346) | 3.096 (0.0332)
  Week 12, hour 4 (n=437, 202, 224) | 3.050 (0.0278) | 2.793 (0.0349) | 3.054 (0.0333)
  Week 12, hour 23, minute 15 (n=430, 200, 214) | 2.991 (0.0282) | 2.799 (0.0349) | 2.985 (0.0341)
  Week 12, hour 23, minute 45 (n=426, 195, 205) | 2.977 (0.0268) | 2.799 (0.0336) | 2.946 (0.0332)
  Week 16, minute 5 (n=429, 207, 218) | 3.016 (0.0301) | 2.753 (0.0362) | 3.009 (0.0355)
  Week 16, minute 15 (n=428, 209, 219) | 3.029 (0.0293) | 2.737 (0.0353) | 3.002 (0.0348)
  Week 16, minute 30 (n=433, 209, 220) | 3.063 (0.0298) | 2.747 (0.0359) | 3.036 (0.0353)
  Week 20, minute 5 (n=430, 206, 218) | 2.985 (0.0286) | 2.744 (0.0349) | 2.966 (0.0338)
  Week 20, minute 15 (n=430, 207, 220) | 3.020 (0.0293) | 2.749 (0.0356) | 2.994 (0.0345)
  Week 20, minute 30 (n=431, 207, 221) | 3.058 (0.0309) | 2.774 (0.0374) | 3.028 (0.0362)
  Week 26, minute 5 (421, 202, 213) | 2.956 (0.0289) | 2.733 (0.0352) | 2.945 (0.0345)
  Week 26, minute 15 (n=414, 200, 207) | 2.980 (0.0298) | 2.713 (0.0363) | 2.959 (0.0360)
  Week 26, minute 30 (n=424, 206, 213) | 2.983 (0.0282) | 2.715 (0.0342) | 2.949 (0.0337)
  Week 26, hour 1 (n=425, 206, 212) | 3.034 (0.0293) | 2.721 (0.0352) | 2.997 (0.0346)
  Week 26, hour 2 (n=420, 203, 208) | 3.049 (0.0308) | 2.777 (0.0370) | 3.036 (0.0366)
  Week 26, hour 3 (n=416, 204, 213) | 3.097 (0.0331) | 2.831 (0.0389) | 3.065 (0.0381)
  Week 26, hour 4 (n=416, 203, 208) | 3.022 (0.0312) | 2.776 (0.0369) | 3.021 (0.0364)
  Week 26, hour 23, minute 15 (n=405, 187, 202) | 2.971 (0.0321) | 2.758 (0.0387) | 2.901 (0.0379)
  Week 26, hour 23, minute 45 (n=401, 185, 198) | 2.952 (0.0305) | 2.759 (0.0373) | 2.883 (0.0368)
  Week 34, minute 5 (n=408, 194, 212) | 2.967 (0.0321) | 2.713 (0.0387) | 2.919 (0.0374)
  Week 34, minute 15 (n=407, 191, 214) | 2.983 (0.0327) | 2.718 (0.0392) | 2.948 (0.0376)
  Week 34, minute 30 (n=410, 196, 215) | 3.002 (0.0333) | 2.690 (0.0400) | 2.947 (0.0386)
  Week 34, hour 1 (n=412, 195, 215) | 3.014 (0.0336) | 2.711 (0.0400) | 2.959 (0.0385)
  Week 42, minute 5 (n=398, 189, 199) | 2.982 (0.0344) | 2.727 (0.0415) | 2.983 (0.0406)
  Week 42, minute 15 (n=405, 188, 201) | 3.001 (0.0336) | 2.713 (0.0410) | 3.001 (0.0398)
  Week 42, minute 30 (n=405, 189, 201) | 3.016 (0.0345) | 2.734 (0.0419) | 3.021 (0.0408)
  Week 50, minute 5 (n=386, 185, 199) | 2.925 (0.0328) | 2.729 (0.0393) | 2.942 (0.0381)
  Week 50, minute 15 (n=391, 187, 203) | 2.971 (0.0330) | 2.729 (0.0398) | 2.962 (0.0384)
  Week 50, minute 30 (n=392, 186, 204) | 2.999 (0.0342) | 2.731 (0.0409) | 2.998 (0.0394)
  Week 52, minute 5 (n=401, 188, 197) | 2.899 (0.0309) | 2.673 (0.0377) | 2.916 (0.0367)
  Week 52, minute 15 (n=394, 183, 200) | 2.942 (0.0314) | 2.701 (0.0389) | 2.969 (0.0371)
  Week 52, minute 30 (n=402, 189, 202) | 2.923 (0.0325) | 2.666 (0.0391) | 2.962 (0.0378)
  Week 52, hour 1 (n=404, 190, 201) | 2.992 (0.0339) | 2.696 (0.0405) | 3.011 (0.0393)
  Week 52, hour 2 (n=402, 186, 202) | 2.997 (0.0354) | 2.727 (0.0421) | 3.005 (0.0405)
  Week 52, hour 3 (n=400, 186, 199) | 3.029 (0.0359) | 2.742 (0.0427) | 3.020 (0.0413)
  Week 52, hour 4 (n=397, 184, 199) | 2.984 (0.0359) | 2.725 (0.0425) | 2.991 (0.0410)
  Week 52, hour 23, minute 15 (n=388, 183, 198) | 2.866 (0.0349) | 2.675 (0.0419) | 2.865 (0.0402)
  Week 52, hour 23, minute 45 (n=395, 185, 199) | 2.869 (0.0342) | 2.694 (0.0406) | 2.868 (0.0390)

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose at Day 1 and Weeks 12, 26, and 52
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 3, and 4 hours post-dose. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: From 5 minutes to 4 hours post-dose at Day 1 and Weeks 12, 26, and 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 519 | 266 | 264
Liters
  Day 1 | 1.570 (0.0075) | 1.373 (0.0092) | 1.514 (0.0092)
  Week 12 (n=460, 214, 232) | 1.560 (0.0134) | 1.384 (0.0170) | 1.531 (0.0164)
  Week 26 (n=430, 206, 216) | 1.546 (0.0160) | 1.369 (0.0194) | 1.495 (0.0190)
  Week 52 (n=405, 192, 203) | 1.502 (0.0162) | 1.336 (0.0203) | 1.487 (0.0196)

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 12 Hours Post-dose at Day 1 and Weeks 12 and 52
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 3, 4, 6, 8 10, and 12 hours post-dose. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: From 5 minutes to 12 hours post-dose at Day 1 and Weeks 12 and 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 144 | 77 | 76
Liters
  Day 1 | 1.566 (0.0168) | 1.407 (0.0207) | 1.534 (0.0206)
  Week 12 (n=133, 69, 70) | 1.539 (0.0261) | 1.398 (0.0324) | 1.505 (0.0320)
  Week 52 (n=125, 62, 58) | 1.492 (0.0265) | 1.364 (0.0352) | 1.424 (0.0344)

14. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 23 Hours 45 Minutes and From 12 Hours to 23 Hours 45 Minutes Post-dose at Weeks 12 and 52
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; 1, 2, 3, 4, 6, 8, 10, and 12 hours; 23 hours 15 minutes; and 23 hours 45 minutes post-dose. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included the same covariates as the primary Outcome Measure.
Time Frame: From 5 minutes to 23 hours 45 minutes post-dose at Weeks 12 and 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 133 | 69 | 70
Liters
  Week 12 | 1.486 (0.0236) | 1.380 (0.0298) | 1.459 (0.0294)
  Week 52 (n=125, 62, 58) | 1.445 (0.0261) | 1.339 (0.0346) | 1.379 (0.0338)

15. Secondary Outcome: Number of Moderate or Severe Exacerbations of Chronic Obstructive Pulmonary Disease (COPD) Per Year During the Study (Baseline to Week 52)
Description: The number of moderate or severe exacerbations of COPD per year during the study was calculated by dividing the total number of exacerbations during the study by the total number of years of treatment. A COPD exacerbation was considered to be moderate if treatment with systemic corticosteroids and/or antibiotic was required. A COPD exacerbation was considered to be severe if treatment for moderate severity and hospitalization was required.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Exacerbations per treatment year
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 525 | 268 | 267
Exacerbations per treatment year | 0.54 [0.496 to 0.869] | 0.80 [0.586 to 1.105] | 0.62 [0.614 to 1.085]

16. Secondary Outcome: Percentage of Patients Who Experienced a Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation During the Study (Baseline to Week 52)
Description: A COPD exacerbation was considered to be moderate if treatment with systemic corticosteroids and/or antibiotic was required. A COPD exacerbation was considered to be severe if treatment for moderate severity and hospitalization was required.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 524 | 266 | 266
Percentage of participants | 32.8 | 40.2 | 30.1

17. Secondary Outcome: Percentage of Nights With "no Nighttime Awakenings" During the Study (Baseline to Week 52)
Description: A night with "no nighttime awakenings" was defined as any night where the patient did not wake up due to 1 or more of 6 symptoms (respiratory symptoms, cough, wheeze, amount of sputum, color of sputum, and breathlessness). Symptoms occurring during the previous 12 hours were recorded each morning and evening by the patient in an electronic diary. The percentage of nights with 'no nighttime awakenings' was calculated as the total number of nights with "no nighttime awakenings" over the 52 week treatment period divided by the total number of nights where diary recordings were made.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 523 | 263 | 262
Percentage of nights | 57.36 (1.842) | 52.15 (2.239) | 55.47 (2.230)

18. Secondary Outcome: Percentage of Days With "no Daytime Symptoms" During the Study (Baseline to Week 52)
Description: A day with "no daytime symptoms" was defined as any day where the patient recorded no cough, no wheeze, no production of sputum, no feeling of breathlessness (other than when running), and no puffs of rescue medication during the previous 12 hours in evening entry in the electronic patient diary. The percentage of days with "no daytime symptoms" was calculated as the total number of days with "no daytime symptoms" over the 52 week treatment period divided by the total number of days where diary recordings were made.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 522 | 263 | 263
Percentage of days | 6.54 (1.208) | 3.81 (1.431) | 7.14 (1.424)

19. Secondary Outcome: Percentage of "Days Able to Perform Usual Daily Activities" During the Study (Baseline to Week 52)
Description: A "day able to perform usual daily activities" was defined as any day where the patient recorded in their electronic diary in the evening that they were not prevented from performing their usual daily activities due to respiratory symptoms during the previous 12 hours. The percentage of "days able to perform usual daily activities" was calculated as the total number of "days able to perform usual daily activities" over the 52 week treatment period divided by the total number of days where diary recordings were made.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 522 | 263 | 263
Percentage of days | 38.02 (1.883) | 36.18 (2.270) | 38.09 (2.259)

20. Secondary Outcome: Change From Baseline in the Mean Daily Total Symptom Score During the Study (Baseline to Week 52)
Description: The daily total symptom score was defined as the sum of the morning and evening patient self-reported diary assessments of 6 symptoms (respiratory symptoms/impact on daily activities, cough, wheeze, amount of sputum, color of sputum, and breathlessness). Means for baseline (14 day maximum run-in period) and the 52 week treatment period were calculated. Mean scores ranged from 0-18, with a higher score indicating worse symptoms. A negative change score indicated improvement.
Time Frame: Baseline to Week 52
Population: Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Number analyzed (Participants) | 523 | 263 | 263
Units on a scale | -1.85 (0.125) | -1.42 (0.149) | -1.87 (0.149)

ADVERSE EVENTS:
Arm/Group | Glycopyrronium Bromide 50 μg | Placebo to Glycopyrronium Bromide | Tiotropium 18 μg
Serious Adverse Events (participants affected / at risk) | 65/525 | 43/268 | 40/267
Other Adverse Events (participants affected / at risk) | 305/525 | 164/268 | 156/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium Bromide 50 μg (N=525) | Placebo to Glycopyrronium Bromide (N=268) | Tiotropium 18 μg (N=267)
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 3
Pyrexia (General disorders) | 0 | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 7 | 4
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pyothorax (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 3 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Renal injury (Renal and urinary disorders) | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Testicular necrosis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 | 16 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium Bromide 50 μg (N=525) | Placebo to Glycopyrronium Bromide (N=268) | Tiotropium 18 μg (N=267)
Diarrhoea (Gastrointestinal disorders) | 10 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 16 | 5 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 6 | 3
Nausea (Gastrointestinal disorders) | 9 | 6 | 4
Oedema peripheral (General disorders) | 9 | 6 | 8
Bronchitis (Infections and infestations) | 19 | 9 | 12
Lower respiratory tract infection (Infections and infestations) | 22 | 9 | 10
Nasopharyngitis (Infections and infestations) | 47 | 15 | 21
Sinusitis (Infections and infestations) | 28 | 14 | 9
Upper respiratory tract infection (Infections and infestations) | 57 | 33 | 29
Upper respiratory tract infection bacterial (Infections and infestations) | 28 | 25 | 20
Urinary tract infection (Infections and infestations) | 14 | 8 | 16
Viral infection (Infections and infestations) | 1 | 6 | 4
Viral upper respiratory tract infection (Infections and infestations) | 9 | 13 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 9 | 12
Dizziness (Nervous system disorders) | 9 | 6 | 5
Headache (Nervous system disorders) | 25 | 14 | 12
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 180 | 106 | 85
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 12 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 4
Hypertension (Vascular disorders) | 20 | 12 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.